CLINICAL TRIAL: NCT01019525
Title: Posture and Pulmonary Function of Mouth-breathing Children
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Waleska da Silveira Venturelli, Universidade Federal do Rio de Janeiro
Other Study IDs: MBPF
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Mouth Breathing
Keywords: respiration; respiratory disorders; Otolaryngology; Otorhinolaryngology; Posture
MeSH Terms: conditions — Mouth Breathing; Respiratory Aspiration; Respiration Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mouth Breathing: Children aged between 8-12 years, with clinical diagnosis of mouth breathing
- Nasal Breathing: Children aged between 8-12 years old, with normal breathing

SUMMARY:
The purpose of this study is to characterize the posture and respiratory function of mouth-breathing children.

DETAILED DESCRIPTION:
Mouth-breathing children presents changes in stomatognathic system, which results in head projection, tension augment in scapular belt muscles and postural adaptations. Although thoracic shape and posture can influence ventilatory dynamics, we didn't find studies addressing pulmonary function of mouth-breathing children. This was a transversal study, designed to analyze the posture of mouth-breathing children, and verify the existence of correlation between posture and pulmonary volumes.

ELIGIBILITY:
Inclusion Criteria:

* Nasal breathing (normal subjects group) or mouth breathing (mouth-breathing group), and the age between eight (08) and twelve (12) for both groups.

Exclusion Criteria:

* Prior physiotherapeutic treatment or in process, presence of diagnostic or report on acute or chronic pulmonary disease, neurofunctional or cognitive impairment and alteration of the osteomuscular system.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mouth-breathing children were referred by Pediatrics Service (Federal University of Rio de Janeiro) and by School of Dentistry (Federal University of Rio de Janeiro), after the diagnosis of mouth breathing was confirmed.
  Nasal breathing children were recruited from Tia Ciata Municipal School (Praça Onze-Rio de Janeiro, Brazil).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary function, by means of forced spirometry. | Within the first 30 days after recruitment.

SECONDARY OUTCOMES:
Posture, by means of photogrammetry. | Within the first 30 days after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara LS Menezes, PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil